CLINICAL TRIAL: NCT03658564
Title: Preoperative Oral Carbohydrate Treatment in Diabetes Patients: A Randomized, Double-blind Trial
Brief Title: Preoperative Oral Carbohydrate Treatment Minimizes Insulin Resistance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: poster2017
Record Dates: First submitted 2018-05-19; First posted 2018-09-05 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-09

CONDITIONS: Insulin Resistance
Keywords: Insulin resistance; Diabetes mellitus; Carbohydrate
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral carbohydrate (Experimental): fast from midnight the night before surgery, and patients consume 400 ml Preoperative oral carbohydrate preOp®(12.5% carbohydrates, 0.5%kcal/ml, 240 mOsm, pH 4.9, Nutricia Zoetermeer, the Netherlands) 3 hours prior to induction of anesthesia and finished the ingestion within 20 minutes.
  Interventions: Dietary Supplement: Preoperative Oral Carbohydrate Drink
- Fasting (No Intervention): fast from midnight the night before surgery, and no preoperative oral carbohydrate loading

INTERVENTIONS:
Dietary Supplement: Preoperative Oral Carbohydrate Drink — Patients in Oral carbohydrate group consumed 400 ml Preoperative Oral Carbohydrate Drink Nutricia preOp® (12.5% carbohydrates, 0.5kcal/ml, 240 mOsm, pH 4.9, Nutricia Zoetermeer, the Netherlands) 3 hours prior to induction of anesthesia and finished the ingestion within 20 minutes.
  Arms: Oral carbohydrate

SUMMARY:
Insulin resistance is a positive protective reaction against surgery .this resistance has some negative consequences for patient health. It is associated with infectious complications. At the same time, Postoperative insulin resistance has been shown to correlate with the length of postoperative stay in hospital. Recently several clinical studies have shown that a carbohydrate-rich drink given 2 h before surgery diminishes postoperative insulin resistance in patient. The aim of our study is to investigate the influence on insulin resistance in patient with diabetes.

DETAILED DESCRIPTION:
Insulin resistance is a positive protective reaction against surgery . As a response to surgery, activation of neuroendocrine and inflammation systems occurs as a protective reaction. However, this resistance has some negative consequences for patient health. It is associated with infectious complications. At the same time, Postoperative insulin resistance has been shown to correlate with the length of postoperative stay in hospital. Recently several clinical studies have shown that a carbohydrate-rich drink given 2 h before surgery diminishes postoperative insulin resistance in patient. The aim of our study is to investigate the influence on insulin resistance in patient with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent elective open colorectal resection for colorectal carcinoma and electric orthopedic surgery

Exclusion Criteria:

* Weight loss greater than 10 per cent during the previous 6 months
* Renal insufficiency (creatinine, > 3 mg/dl; hemodialysis)
* Hepatic insufficiency (Child-Pugh class, ≥ B)
* Gastro-oesophageal reflux disease
* Gastrointestinal obstruction or conditions (including pharmacological treatment) known to affect gastric emptying rate

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-09-30 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
VAS | 1 day (preoperative period)
  Preoperative general well-beings before assessed with the visual analogue scale (VAS).

SECONDARY OUTCOMES:
HOMA | perioperative period)
  Preoperative insulin resistance before and immediately after the surgery assessed with the homeostasis model assessment (HOMA)

CONTACTS AND LOCATIONS:
Overall Officials: yang z Xiao, MD,PhD, Study Director — 0866-17709873399
Locations (1):
- The Second Hospital of Dalian Medical University, Dalian, Liaoning, China